CLINICAL TRIAL: NCT02211313
Title: Evaluation of Ureteral Stents in the Management of Stone Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of further funding.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201205184
Record Dates: First submitted 2014-08-04; First posted 2014-08-07 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Urinary Stones; Urinary Tract Stones
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ureteral stent - soft, 6 French (Active Comparator): Subjects randomized to soft stent, size 6 French
  Interventions: Device: Randomization to size 6 French soft vs. size 6 French hydrophobic ureteral stent.
- Ureteral stent - hydrophobic, 6 French (Active Comparator): Subjects randomized to hydrophobic stent, size 6 French
  Interventions: Device: Randomization to size 6 French soft vs. size 6 French hydrophobic ureteral stent.

INTERVENTIONS:
Device: Randomization to size 6 French soft vs. size 6 French hydrophobic ureteral stent. — Subjects will be randomized to one of two study arms according to ureteral stent size and degree of firmness (size 6Fr, soft vs. size 6Fr, hydrophobic) with allocation ratio of 1:1.

SUMMARY:
A thin tube, called a ureteral stent, is inserted into the ureter and is commonly used as treatment of urinary stone disease. Stents are designed to help provide drainage of the kidney in the setting of an obstructing stone, or postoperative swelling of the ureter. Though their presence is only temporary, stents are associated with a significant amount of patient discomfort and bother, which can negatively impact overall satisfaction. Over the past decades, there have been refinements in stent technology and usage philosophy. Smaller and softer stents are now available for use in patients, though studies evaluating the relative benefits have been conflicting. The investigators aim to evaluate the effect of stent size and composition upon outcomes after the treatment of stone disease, including patient comfort and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age and willing and able to provide informed consent
2. Patients with current urinary stone disease, undergoing any of the following procedures:

   * cystoscopy with stent placement
   * ureteroscopy with intracorporeal lithotripsy

Exclusion Criteria:

1. Patients with compromised urinary tract due to cancer (e.g. bladder tumor, ureteral obstruction from non-GU malignancy)
2. Patients requiring bilateral surgical stone management procedure
3. Patients with any single stone exceeding 1.5 cm
4. Patients with severe concurrent disease, infection, or co-morbidity that, in the judgment of the investigator, would render the patient inappropriate for enrollment
5. Any patient who is on anticholinergic medication at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-08; Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alana C Desai, M.D., Principal Investigator — Washington UniversitySchool of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ureteral Stent - Soft, 6 French | Ureteral Stent - Hydrophobic, 6 French
Started | 18 | 23
Completed | 12 | 20
Not Completed | 6 | 3
Not completed — Treatment Failure | 5 | 2
Not completed — No Follow up Questionnaires | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ureteral Stent - Soft, 6 French | Ureteral Stent - Hydrophobic, 6 French | Total
Number analyzed (Participants) | 18 | 23 | 41
Age, Categorical [Count of Participants; unit: Participants] — Population: 5 soft and 2 hydrophobic patients failed treatment. 1 soft and 1 hydrophobic patients have no follow up questionnaires.
  Participants
    number analyzed (Participants) | 12 | 20 | 32
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 6 | 15 | 21
    >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 5 soft and 2 hydrophobic patients failed treatment. 1 soft and 1 hydrophobic patients have no follow up questionnaires.
  Participants
    number analyzed (Participants) | 12 | 20 | 32
    Female | 6 | 13 | 19
    Male | 6 | 7 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 5 soft and 2 hydrophobic patients failed treatment. 1 soft and 1 hydrophobic patients have no follow up questionnaires.
  Participants
    Race: number analyzed (Participants) | 12 | 20 | 32
    Race: African American | 0 | 3 | 3
    Race: Caucasian | 12 | 17 | 29
Region of Enrollment [Count of Participants; unit: Participants] — Population: 5 soft and 2 hydrophobic patients failed treatment. 1 soft and 1 hydrophobic patients have no follow up questionnaires.
  Participants
    United States: number analyzed (Participants) | 12 | 20 | 32
    United States | 12 | 20 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain on the 10-point Analog Pain Scale at Day 7 Post Stent Removal.
Description: The 10-point scale ranges from 0 (zero) for no pain (minimum) to 10 for the worst possible pain (maximum). The unit of measure is 1 point on the 10-point scale.
Time Frame: Baseline, day 7 post stent removal
Measure: Mean (Standard Deviation); unit: Scores on a scale 0-10 (Numeric)
Arm/Group | Ureteral Stent - Soft, 6 French | Ureteral Stent - Hydrophobic, 6 French
Number analyzed (Participants) | 12 | 20
Scores on a scale 0-10 (Numeric)
  Pre Stent: Pain rating 0-10 (Numeric) | 1.3 (1.7) | 1.5 (2.3)
  In-Situ: Pain rating 0-10 (Numeric) | 4.0 (3.5) | 4.8 (3.4)
  Post: Pain rating 0-10 (Numeric) | 0.7 (1.1) | 1.1 (2.1)

ADVERSE EVENTS:
Time Frame: From the time of the initial stent placement through the completion of the 7 day post stent removal questionnaires. The timeframe in which data was collected for adverse events was up to 27 days.
Description: Participation in the study did not pose any risks to the participants beyond what was expected from the standard of care surgical stone management procedure.
Arm/Group | Ureteral Stent - Soft, 6 French | Ureteral Stent - Hydrophobic, 6 French
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/20
Other Adverse Events (participants affected / at risk) | 0/12 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT02211313/Prot_SAP_000.pdf